CLINICAL TRIAL: NCT04066439
Title: The Marker Expression of Corneal Surface From Penetrating Keratopathy After Collagenase A Assisted COMET Case Series
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201905046RINC
Record Dates: First submitted 2019-08-15; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cornea biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: specimen — Immunohistochemistry analysis

SUMMARY:
In order to examine the cells of the corneal epithelium in the patients who receive corneal transplantation after collagenase A assisted cultivated oral mucosa epithelium transplant (CA-COMET), we analyzed the specimens from penetrating keratoplasty with immunochemical staining.

DETAILED DESCRIPTION:
Limbal insufficiency may cause persistent corneal erosion, turbidity, and even infection and blindness, leading to major eye damage. In patients with limbal stem cell insufficiency, due to the defect of the limbal stem cells, the new epidermal cells cannot be produced, and without the limbus as a barrier, the cells near the conjunctiva will move toward the center of the cornea, result in replacing the corneal cells and causing corneal conjunctivalization.

In recent years, many surgical methods for treating corneal stem cell defects include amniotic membrane transplantation, autologous limbal cell transplantation, and allogeneic limbal cell transplantation. However, in patients with bilateral total limbal insufficiency, there are no autologous limbal cells in the contralateral eye, and allografts may also have rejection and infection.

Cultured oral mucosa epithelium transplant is a method for treating bilateral full-limbal cell defects. The patient's own oral mucosal cells are cultured in the laboratory, and the cultured epithelium is transplanted to the patient's limbus. In the experiment, mouse cells are used as a feeder cell and transplanted to the human body, which is prone to potential problems such as rejection or infection. In order to resolve these problems, our laboratory modified the process of separating the limbal stem cells. By replacing the dispase II/trypsin-EDTA with Collagenase A, there were no needs to use a feeder cell. This experiment has been successfully completed under the national plan.

In this study, we want to investigate the cells on the ocular surface form the four patients who underwent corneal transplantation after receiving CA-COMET.

Dr.Kuan-Ting Kuo, a pathologist in NTUH, will assist us in the staining of the specimens of the cornea from four patients who underwent corneal transplantation after receiving CA-COMET. The specimens of the four patients will be stained (Immunohistochemistry) with markers of the cornea and conjunctival cells (K3, K4, K12, K13, K19, MUC5, P63).

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent corneal transplantation after receiving CA-COMET in five years.

Exclusion Criteria:

* The patients who NEVER underwent corneal transplantation after receiving CA-COMET.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent corneal transplantation after receiving CA-COMET in five years.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-06 (Estimated); Study Completion 2020-08-06 (Estimated)

PRIMARY OUTCOMES:
Immunofluorescence staining | 1 year
  Using fluorescence microscope to detect specific biomolecule targets with markers of the cornea and conjunctival cells (K3, K4, K12, K13, K19, MUC5, P63)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan